CLINICAL TRIAL: NCT05315609
Title: Effects of Virtual Reality Meditation in Older Adults: A Randomized Controlled Trial
Brief Title: Effects of Virtual Reality Meditation in Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lady Davis Institute (Other)
Responsible Party: Principal Investigator, Soham Rej MD, MSc, Primary Investigator, Lady Davis Institute
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IUSMD-21-48
Record Dates: First submitted 2021-08-11; First posted 2022-04-07 (Actual); Last update posted 2025-06-11 (Actual); Status verified 2022-03

CONDITIONS: Older Adults; Stress; Mental Disorder
Keywords: Virtual reality; Meditation; Mindfulness; Stress; Older adults
MeSH Terms: conditions — Mental Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention: Virtual Reality Mindfulness Group (Experimental): The intervention will be 4-weeks, twice per week, 15-minute/session VR-mindfulness intervention group.
  Interventions: Behavioral: VR Meditation
- No intervention: Waitlist Control Group (No Intervention): These participants will be on a waitlist to receive the VR guided meditation program after data collection has been completed (after the 4 weeks)

INTERVENTIONS:
Behavioral: VR Meditation — This 4-week VR program will use the Oculus Pro-Quest 2 headsets for the 15-minute seated VR meditation twice per week for a total of 8 sessions over the 4 weeks.
  Arms: Intervention: Virtual Reality Mindfulness Group

SUMMARY:
Virtual reality (VR) allows users to interact within a simulated environment using electronic devices such as a VR headset or goggles. Multiple studies with younger adults have demonstrated that VR meditation can be an important tool in reducing stress, however, this has not been studied in older adults. In this study, the investigators aim to assess the effects of a 4-week program of 15-minutes sessions, twice per week of meditation delivered through VR with the aim of evaluating its impact on stress in older adults.

ELIGIBILITY:
Inclusion Criteria:

* Living in the Greater Montreal area and able to speak English or French
* Perceived Stress Score (PSS)equal or greater than 10
* Over >=60 years of age

Exclusion Criteria:

* Diagnosis of epilepsy, schizophrenia, brain tumor
* History of recurrent migraines or seizures or TBI in the past year
* Substance use disorders in the last year
* Psychiatric hospitalizations in the last year.
* Acute psychotic symptoms
* Acute suicidal ideation or intent
* Glaucoma
* PTSD
* Changes to psychoactive medications in the past 4 weeks
* Alcohol, caffeine or cannabis consumption within 24 hr before the session, or nicotine consumption within 15 min of the session
* Important hearing impairment
* Recovery phase of any eye surgery

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2022-04-30 (Actual); Primary Completion 2022-05-01 (Actual); Study Completion 2022-09-01 (Actual)

PRIMARY OUTCOMES:
Changes in stress scores as measured by the Perceived Stress Scale (PSS) for treatment group versus control group | Baseline, Once weekly during intervention
  To assess the effectiveness of the virtual reality meditation program in reducing stress in older adults.
  Scores on the PSS can range from 0-40, with higher scores indicating higher perceived stress.

SECONDARY OUTCOMES:
Changes in symptoms of anxiety as measured by the Generalized Anxiety Disorder-7 (GAD-7) questionnaire for treatment group versus control group | Baseline, Once weekly during intervention
  To assess the effects of the virtual reality meditation program on symptoms of anxiety in older adults.
  Scores on the GAD-7 range from 0-21, with higher scores indicating more severe anxiety.
Changes in symptoms of depression as measured by the Patient Health Questionnaire-9 (PHQ-9) scale for treatment group versus control group | Baseline, Once weekly during intervention
  To assess the effects of the virtual reality meditation program on symptoms of depression in older adults.
  Scores on the PHQ-9 can range from 0-27, with higher scores indicating more severe depression.

OTHER OUTCOMES:
Changes in symptoms of mindfulness skills | Baseline, Once weekly during intervention
  To assess the effects of the virtual reality meditation program on mindfulness skills in older adults.
  Facet Mindfulness Questionnaire - Short Form (FFMQ-SF) is a 24-item scale that is used to assess whether mindfulness is related to a decrease in clinical symptoms of depression, anxiety, and stress.
Qualitative Component: Participant observation, semi-structured interviews, and a focus group with participants. | Post intervention (4-weeks)
  Qualitative interviews to examine users' experience of the virtual reality meditation program.
  We will conduct qualitative evaluations through participant observation and semi-structured interviews and a focus group with participants. The qualitative part of the study will analyze service users' experience, engagement, and challenges throughout the study. Participant observation will be used to provide a context for the interviews. It will also help to observe clients' engagement, usage, expressions, physical movements, and barriers.
Changes in simulator sickness as measured by the Simulator Sickness Questionnaire | Baseline, Once weekly during intervention
  To assess participants' acceptability of the virtual reality guided meditation program.
  Simulator Sickness Questionnaire is a 16-item scale that is widely used to assess simulator sickness.
Changes in loneliness sentiments as measured by the University of California-3 (UCLA-3) item loneliness questionnaire | Baseline, Once weekly during intervention
  To assess the effects of the virtual reality meditation program on feelings of loneliness measured through the University of California-3 (UCLA 3-item) loneliness scale.
  The Three-Item Loneliness Scale is an interviewer-administered questionnaire developed from the Revised UCLA Loneliness Scale. Each question is rated on a 3-point scale: 1 = Hardly Ever; 2 = Some of the Time; 3 = Often. All items are summed to give a total score.
  Higher scores indicate greater feelings of loneliness
Changes in symptoms of sleep quality as measured by the Athens Insomnia Scale (AIS) | Baseline, Once weekly during intervention
  To assess the effects of the virtual reality meditation program on sleep quality in older adults.
  Each item is rated on a 4-point numerical rating scale (NRS; where 0= no problem at all and 3= very serious problem). Total scores range from 0 to 24 in the AIS-8 and from 0 to 15 in the AIS-5. Higher scores in these AIS measures indicate that responders have severe insomnia symptoms.
Changes in symptoms of quality of life in older adults as measured by the European Quality of Life (Euro-QoL) measure. | Baseline, Once weekly during intervention
  To assess the effects of the virtual reality meditation program on quality of life in older adults.
  Descriptive data from the 5 dimensions of Part I can be used to generate a health-related quality of life profile for the subject. Part II is scored from 0 (worst health state imaginable) to 100 (best health state imaginable). The score from Part II can be used to track changes in health, on an individual or group level, over time (McDowell & Newell, 1996).
Changes in sense of presence as measured by the ITC-Sense of Presence Inventory | Baseline, Once weekly during intervention
  The ITC-Sense of Presence Inventory is a self-report presence measure to evaluate experiential aspects of immersive technology.

CONTACTS AND LOCATIONS:
Locations (2):
- Canada (2):
  - Douglas Mental Health University Institute, Montreal, Quebec
  - Lady Davis Institute/ Jewish General Hospital, Montreal

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cinalioglu K, Lavin P, Bein M, Lesage M, Gruber J, Se J, Bukhari S, Sasi N, Noble H, Andree-Bruneau M, Launay C, Sanders J, Gauthier S, Rosa P, Lifshitz M, Battistini BJ, Beauchet O, Khoury B, Bouchard S, Fallavollita P, Vahia I, Rej S, Sekhon H. Effects of virtual reality guided meditation in older adults: the protocol of a pilot randomized controlled trial. Front Psychol. 2023 Jul 28;14:1083219. doi: 10.3389/fpsyg.2023.1083219. eCollection 2023. PMID 37575420